CLINICAL TRIAL: NCT05891886
Title: Supplemental Oxygen in Pulmonary Embolism (SO-PE)
Acronym: SO-PE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Christopher Kabrhel MD MPH, Professor of Emergency Medicine; Attending Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2023P000252
Record Dates: First submitted 2023-05-04; First posted 2023-06-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism; Metabolomics; Oxygen Inhalation Therapy
Keywords: Pulmonary Embolism; PE; Right ventricular dysfunction
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism; Ventricular Dysfunction, Right | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Supplemental oxygen delivered by facemask (Experimental): Patients with acute PE will be randomized to breathing supplemental oxygen by non-rebreather face mask first.
  Subjects will alternate treatments (supplemental oxygen or room air) every 30 minutes for 90 minutes (e.g. T=30, T=60, T=90) and then will maintain their treatment (oxygen or room air) for a total of 180 minutes.
  Interventions: Drug: Oxygen Therapy; Device: Non-rebreather mask
- Room air delivered by facemask (Active Comparator): Patients with acute PE will be randomized to breathing room air by non-rebreather face mask first.
  Subjects will alternate treatments (supplemental oxygen or room air) every 30 minutes for 90 minutes (e.g. T=30, T=60, T=90) and then will maintain their treatment (oxygen or room air) for a total of 180 minutes.
  Interventions: Device: Non-rebreather mask

INTERVENTIONS:
Drug: Oxygen Therapy — Study subjects will be asked to breathe supplemental, or extra, oxygen during several time periods.
  Arms: Supplemental oxygen delivered by facemask
Device: Non-rebreather mask — Non-rebreather mask is a non-invasive oxygen supplementation device that is used to provide continuous oxygen flow, typically in a hospital setting.
  Other Names: NRM (Non-rebreather mask)

SUMMARY:
A study of how supplemental oxygen helps patients with acute pulmonary embolism (PE).

Hypothesis: Oxygen affects right ventricular dysfunction (RVD) in patients with acute pulmonary embolism (PE) primarily by relieving hypoxic pulmonary vasoconstriction and reducing pulmonary pressure (PA) pressure, and that this process is metabolically driven.

DETAILED DESCRIPTION:
In the Emergency Department (ED), investigators will perform a randomized, crossover trial of adult patients with acute PE.

Study subjects will be randomized to one of two interventions (supplemental oxygen delivered by facemask) vs. room air. Therapy will be alternated at t=30, t=60, t=90 minutes, and then maintained for 180 minutes.

After each treatment change, and at 180 minutes, investigators will: 1) perform echocardiograms to determine how oxygen affects right ventricular dysfunction (RVD) and, 2) draw blood for metabolomic analyses to determine the metabolic pathways that change in response to oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Confirmed Pulmonary Embolism (PE) on imaging <24 hours prior to enrollment
* New symptom onset and / or worsening symptoms <72 hours
* Confirmation of right ventricular dysfunction (RVD) by clinician
* Oxygen saturation ≥90% while breathing room air

Exclusion Criteria:

* Hemodynamic instability
* Use of vasopressors or mechanical circulatory support
* Planned use of thrombolytics or plan for embolectomy
* Oxygen saturation <90% while breathing room air
* New onset arrhythmia
* History of pulmonary hypertension, severe chronic obstructive pulmonary disease (COPD) requiring home oxygen or chronic steroid use, hypoventilation syndrome requiring continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), or congestive heart failure (CHF) with LV ejection fraction < 40% or chronic oxygen therapy
* Known pregnancy
* Vasodilator medication used in the past 24 hours
* Symptom onset ≥72 hours
* Inability to wear a face mask
* Inability to obtain adequate baseline echocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery systolic pressure (PASP) | 30 minutes after study treatment (supplemental oxygen) or placebo (room air)
  PASP is measured on bedside echocardiogram
Pulmonary artery systolic pressure (PASP) | 60 minutes after study treatment (supplemental oxygen) or placebo (room air)
  PASP is measured on bedside echocardiogram
Pulmonary artery systolic pressure (PASP) | 90 minutes after study treatment (supplemental oxygen) or placebo (room air)
  PASP is measured on bedside echocardiogram
Pulmonary artery systolic pressure (PASP) | 180 minutes after study treatment (supplemental oxygen) or placebo (room air)
  PASP is measured on bedside echocardiogram

SECONDARY OUTCOMES:
Right ventricular to left ventricular ratio (RV/LV) | 30 minutes after study treatment (supplemental oxygen) or placebo (room air)
  RV/LV ratio is measured on bedside echocardiogram
Right ventricular to left ventricular ratio (RV/LV) | 60 minutes after study treatment (supplemental oxygen) or placebo (room air)
  RV/LV ratio is measured on bedside echocardiogram
Right ventricular to left ventricular ratio (RV/LV) | 90 minutes after study treatment (supplemental oxygen) or placebo (room air)
  RV/LV ratio is measured on bedside echocardiogram
Right ventricular to left ventricular ratio (RV/LV) | 180 minutes after study treatment (supplemental oxygen) or placebo (room air)
  RV/LV ratio is measured on bedside echocardiogram
Concentrations of circulating metabolites and metabolic profiles measured by high-throughput metabolomic assays | 30 minutes after study treatment (supplemental oxygen) or placebo (room air)
  Investigators will perform high-throughput metabolomics to identify changes in circulating blood metabolites associated with supplemental oxygen use in patients with acute PE.
Concentrations of circulating metabolites and metabolic profiles measured by high-throughput metabolomic assays | 60 minutes after study treatment (supplemental oxygen) or placebo (room air)
  Investigators will perform high-throughput metabolomics to identify changes in circulating blood metabolites associated with supplemental oxygen use in patients with acute PE.
Concentrations of circulating metabolites and metabolic profiles measured by high-throughput metabolomic assays | 90 minutes after study treatment (supplemental oxygen) or placebo (room air)
  Investigators will perform high-throughput metabolomics to identify changes in circulating blood metabolites associated with supplemental oxygen use in patients with acute PE.
Concentrations of circulating metabolites and metabolic profiles measured by high-throughput metabolomic assays | 180 minutes after study treatment (supplemental oxygen) or placebo (room air)
  Investigators will perform high-throughput metabolomics to identify changes in circulating blood metabolites associated with supplemental oxygen use in patients with acute PE.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kabrhel, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.
  The results of this study will be published in scientific journals and presented at national/international scientific meetings.

REFERENCES:
- [Derived] Lyhne MD, Liteplo AS, Zeleznik OA, Dudzinski DM, Andersen A, Shokoohi H, Al Jalbout N, Eke OF, Morone CC, Huang CK, Heyne TF, Kalra MK, Kabrhel C. Supplemental oxygen for pulmonary embolism (SO-PE): study protocol for a mechanistic, randomised, blinded, cross-over study. BMJ Open. 2024 Nov 12;14(11):e091567. doi: 10.1136/bmjopen-2024-091567. PMID 39532350